CLINICAL TRIAL: NCT00003802
Title: A Phase II Trial of Pyrazoloacridine (NSC 366140, IND 36325) in Metastatic Cutaneous and Ocular Melanoma
Brief Title: Pyrazoloacridine in Treating Patients With Metastatic Skin or Eye Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: JHOC-J9875, CDR0000066946; U01CA063437 (NIH); P30CA006973 (NIH); JHOC-98111005; JHOC-JH9875; JHOC-T96-0116; NCI-T96-0116
Record Dates: First submitted 1999-11-01; First posted 2003-05-02 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — NSC 366140

INTERVENTIONS:
Drug: pyrazoloacridine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of pyrazoloacridine in treating patients who have metastatic skin or eye melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the antitumor activity of pyrazoloacridine (PZA) in chemotherapy naive patients with metastatic cutaneous or ocular melanoma.
* Determine the toxic effects of PZA in this patient population.
* Determine the pharmacokinetic profile of PZA in these patients.

OUTLINE: Patients are stratified into cutaneous or ocular melanoma treatment groups.

Patients receive pyrazoloacridine IV over 3 hours on day 1. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 28-70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic cutaneous or ocular melanoma that is chemotherapy naive
* Bidimensionally measurable disease
* No pleural effusions or ascites
* No untreated CNS metastases
* Stable brain metastases by CT or MRI scan

  * At least 4 weeks since prior steroid therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 4,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN (unless due to hepatic metastases)

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active infection
* No known hypersensitivity to E.coli derived proteins
* No other serious medical problems
* No more than 1 primary malignancy within past 5 years, other than:

  * Nonmelanomatous skin cancer
  * Carcinoma in situ of the cervix
* No history of spinal cord compression

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed (e.g., interleukin-2, interferon alfa, or vaccine therapy)

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Prior radiotherapy for primary ocular melanoma, brain metastases, or to metastatic sites encompassing less than 25% of the bone marrow allowed
* No other prior radiotherapy

Surgery:

* At least 2 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H. Sharfman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States